CLINICAL TRIAL: NCT01941004
Title: A 12 Month Study, With a 6-month, Double-blind, Randomized, Placebo-controlled, Multi-center Parallel- Groups, Treatment Phase Evaluating Efficacy and Safety of Fingolimod 0.5 mg and a 6-month, Open-label, Treatment Phase, in Chinese Patients With Relapsing-remitting Multiple Sclerosis
Brief Title: Safety and Efficacy of Fingolimod in MS Patients in China
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CFTY720D2315
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Multiple Sclerosis (Relapsing Remitting)
Keywords: multiple sclerosis (MS); relapsing remitting multiple sclerosis (RRMS); fingolimod
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- double blinded Fingolimod 6 mos + open label fingolimod 6 mos (Experimental): Randomized to 6 month (180 days) 0.5 mg fingolimod + 6 month (180 day) open label 0.5mg fingolimod capsules for oral administration once daily
  Interventions: Drug: fingolimod
- Placebo 6 mos + open label fingolimod 6 mos (Placebo Comparator): Randomized to 6 month (180 days) matching placebo + 6 month (180 day) open label 0.5mg fingolimod capsules for oral administration once daily
  Interventions: Drug: Placebo (6mos) + open label fingolimod (6 mos)

INTERVENTIONS:
Drug: fingolimod — Randomized to 6 month (180 days) 0.5 mg fingolimod + 6 month (180 day) open label 0.5mg fingolimod capsules for oral administration once daily
  Arms: double blinded Fingolimod 6 mos + open label fingolimod 6 mos
Drug: Placebo (6mos) + open label fingolimod (6 mos) — Randomized to 6 month (180 days) matching placebo + 6 month (180 day) open label 0.5mg fingolimod capsules for oral administration once daily
  Arms: Placebo 6 mos + open label fingolimod 6 mos

SUMMARY:
To evaluate the safety and efficacy of fingolimod 0.5mg vs. placebo in MS patients in China

ELIGIBILITY:
Inclusion Criteria:

-Patients must have relapsing remitting multiple sclerosis

Exclusion Criteria:

Patients with:

* History of chronic immune disease
* Certain cancers
* Uncontrolled diabetes
* Certain eye disorders -Negative for varicella
* zoster virus IgG antibodies
* Certain hepatic conditions
* Low white blood cell count
* On certain immunosuppressive medications or heart medications
* Certain heart conditions or certain lung conditions
* Inability to undergo MRI scans -Diagnosis of Neuromyelitis optica.
* Other protocol defined inclusion/exclusion criteria may apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
number of new/newly enlarged T2 MRI lesions over 6 months | 6 months
  Cumulative number of new/newly enlarged T2 lesions over 6 months

SECONDARY OUTCOMES:
annualized relapse rate (ARR) | 6 months
  The annualized relapse rate (ARR) is identified as the average number of confirmed relapses per year (the total number of confirmed relapses divided by the total days in the study multiplied by 365.25). The number of relapses will include all the confirmed relapses during the study. The time spent in the study will correspond to the observation period for all the relapses from first dose on the study drug to end of study.
number of Gd-enhancing T1 lesions | 6 months
Safety and tolerability of fingolimod 0.5 mg compared to placebo | 12 months
  Based on frequency of adverse events (the number and percentage of patients having any AE by primary system organ class and preferred term) and on the incidence of clinically notable abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals